CLINICAL TRIAL: NCT03396380
Title: Effect of Adding Vitamin D Supplement to Clomiphene Citrate for Induction of Ovulation in Overweight Women With Polycystic Ovary Syndrome
Brief Title: Effect of Vitamin D Supplement in Induction of Ovulation in Overweight Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ain shams maternity hospital
Record Dates: First submitted 2017-12-16; First posted 2018-01-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Ovulation Induction
MeSH Terms: interventions — Vitamin D; Calcium; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin D (Active Comparator): 93 women who will receive clomiphene citrate for induction of ovulation with vitamin D and calcium supplement
  Interventions: Drug: Vitamin D with calcium and clomiphene citrate
- placebo (Placebo Comparator): 93 women who will receive clomiphene citrate for induction of ovulation with placebo and calcium supplement
  Interventions: Drug: Placebo Oral Tablet with calcium and clomiphene citrate

INTERVENTIONS:
Drug: Vitamin D with calcium and clomiphene citrate — 1. Vitamin D ( ossofortin®, EVA PHARMA) 10000 IU twice weekly and calcium (calciprex®, Marcyrl Pharmaceutical Industries ) 1250 mg twice daily which provide elemental calcium 500 mg/tablet for one month before induction of ovulation and both will be continued during the 3 induction cycles in the same regimen.
  2. Induction of ovulation by clomiphene citrate (Clomid®, Aventis) 50 mg tablet twice daily 12 hours apart (total dose 100 mg daily) starting from the third day of menstrual cycle and for five days .
  Arms: vitamin D
Drug: Placebo Oral Tablet with calcium and clomiphene citrate — 1. The placebo tablet twice weekly and calcium (calciprex®, Marcyrl Pharmaceutical Industries ) 1250 mg twice daily which provide elemental calcium 500 mg/tablet for one month before induction of ovulation and both will be continued during the 3 induction cycles in the same regimen.
  2. induction of ovulation by clomiphene citrate (Clomid®, Aventis) 50 mg tablet twice daily 12 hours apart (total dose 100 mg daily)starting from the 3rd day of menstrual cycle and for five days
  Arms: placebo

SUMMARY:
The aim of this work is to evaluate the effect of vitamin D supplementation in overweight infertile women with PCOs undergoing induction of ovulation.

DETAILED DESCRIPTION:
The study will include overweight infertile women with PCOS seeking fertility who will receive induction of ovulation by clomiphene citrate will be recruited and randomized into two groups:

Group A (study group): 93 women who will receive clomiphene citrate for induction of ovulation with vitamin D and calcium supplement

Group B (control group): 93 women who will receive clomiphene citrate for induction of ovulation with placebo and calcium supplement

ELIGIBILITY:
Inclusion Criteria:

* polycystic ovarian syndrome diagnosis made according to ESHRE/ASRM criteria.
* infertility is the cause for seeking treatment.
* overweight females with BMI more than 25 but less than 30.

Exclusion Criteria:

* causes of infertility other than PCOS.
* causes of anovulation other than PCOS.
* current or in last six months use of hormonal treatment.
* contraindication to any drug used in the study.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of ovulation | till cycle day 21 if not reaching more than 18 mm
  * Transvaginal ultrasound will be done to detect signs of ovulation: corpus luteum, fluid in cul-de-sac, collapse of the follicle size.
  * Serum progesterone will be measured in the mid luteal day of the cycle, where:
  Level 19 nmol/L indicates Ovulation. Level <5 nmol/L suggests Ovulation did not occur

SECONDARY OUTCOMES:
Number of growing follicles. | till cycle day 21 if not reaching more than 18 mm
  to monitor induction
Evaluation of the endometrial thickness | in cycle day 14 and 21.
  could be impaired with antiestrogenic effect of clomiphen citrate
Pregnancy rates | pregnancy test 1 week after missed menses
  both clinical and biochemical
Adverse effects | for 3 months
  hot flashes, headache, nausea, vomiting, breast tenderness, blurred vision, abdominal distention and pain and ovarian enlargement or hyperstimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Abbassya, Egypt

REFERENCES:
- [Derived] Rasheedy R, Sammour H, Elkholy A, Salim Y. The efficacy of vitamin D combined with clomiphene citrate in ovulation induction in overweight women with polycystic ovary syndrome: a double blind, randomized clinical trial. Endocrine. 2020 Aug;69(2):393-401. doi: 10.1007/s12020-020-02315-3. Epub 2020 May 3. PMID 32363556